CLINICAL TRIAL: NCT04220450
Title: T1-mapping by Cardiovascular Magnetic Resonance Imaging to Assess Non-Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Andreas Kammerlander (Other)
Responsible Party: Sponsor-Investigator, Dr. Andreas Kammerlander, Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: NAFLD-CMR-2436
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: NAFLD; Heart Failure; Valvular Disease; Coronary Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Heart Failure; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: T1 mapping on Cardiovascular Magnetic Resonance Studies — On clinically indicated Cardiovascular Magnetic Resonance Imaging Studies, native T1-times and extracellular volume will be determined

SUMMARY:
On clinically indicated Cardiovascular Magnetic Resonance studies, native T1-times and extracellular volume of the liver will be assessed and findings correlated with established risk calculators for non-alcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Referred for Cardiovascular Magnetic Resonance Imaging

Exclusion Criteria:

* Non-compatible Devices

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All-comer cohort referred for Cardiovascular Magnetic Resonance Imaging
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Correlation NAFLD and liver T1mapping | cross-sectional within one year
  Correlation NAFLD risk score and liver T1-mapping (native and ECV9

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mascherbauer K, Dona C, Koschutnik M, Dannenberg V, Nitsche C, Duca F, Heitzinger G, Halavina K, Steinacher E, Kronberger C, Bardach C, Beitzke D, Loewe C, Waldmann E, Trauner M, Barkto P, Goliasch G, Mascherbauer J, Hengstenberg C, Kammerlander A. Hepatic T1-Time Predicts Cardiovascular Risk in All-Comers Referred for Cardiovascular Magnetic Resonance: A Post-Hoc Analysis. Circ Cardiovasc Imaging. 2022 Oct;15(10):e014716. doi: 10.1161/CIRCIMAGING.122.014716. Epub 2022 Oct 18. PMID 36256728